CLINICAL TRIAL: NCT00568022
Title: A Phase I Study of Ixabepilone in Combination With Capecitabine in Japanese Patients With Metastatic Breast Cancer Previously Treated With an Anthracycline and a Taxane
Brief Title: A Phase I Study of Ixabepilone in Combination With Capecitabine in Japanese Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA163-117
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ixabepilone; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ixabepilone + Capecitabine (Experimental)
  Interventions: Drug: Ixabepilone; Drug: Capecitabine

INTERVENTIONS:
Drug: Ixabepilone — Ixabepilone: Intravenous (IV) Solution, IV, 32(40)mg/m^2, once every 3 weeks, up to 6 cycles
  Other Names: IXEMPRA; BMS-247550
Drug: Capecitabine — Capecitabine: Tablets, Oral, 1650(2000)mg/m^2, twice daily for 2 weeks, one week off, up to 6 cycles

SUMMARY:
The purpose of this study is to determine the dose-limiting toxicity (DLT), maximum tolerated dose (MTD) and recommended Phase II dose of ixabepilone in combination with capecitabine in Japanese participants with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 20 years
* Histologically or cytologically confirmed diagnosis of adenocarcinoma originating in the breast

Exclusion Criteria:

* Number of prior chemotherapy lines of treatment in the metastatic setting ≥3

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- Japan (4):
  - Local Institution, Matsuyama, Ehime
  - Local Institution, Maebashi, Gunma
  - Local Institution, Osaka, Osaka
  - Local Institution, Sunto-Gun, Shizuoka

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 4 sites in Japan.
Groups:
- Ixabepilone 32 mg/m^2 + Capecitabine 1650 mg/m^2/Day: Ixabepilone 32 mg/m^2 was administered via intravenous (IV) infusion over 3 hours on Day 1 of each 21-day treatment cycle. Capecitabine 1650 mg/m^2/day was administered on Days 1 to 14 of each 21-day treatment cycle.
- Ixabepilone 40 mg/m^2 + Capecitabine 1650 mg/m^2/Day: After receiving Ixabepilone 32 mg/m^2 + Capecitabine 1650 mg/m^2/Day, the dose was escalated such that participants received Ixabepilone 40 mg/m^2 administered via intravenous (IV) infusion over 3 hours on Day 1 of each 21-day treatment cycle. Capecitabine 1650 mg/m^2/day was administered on Days 1 to 14 of each 21-day treatment cycle.
- Ixabepilone 40 mg/m^2 + Capecitabine 2000 mg/m^2/Day: After receiving Ixabepilone 40 mg/m^2 + Capecitabine 1650 mg/m^2/Day, the dose was escalated such that participants received Ixabepilone 40 mg/m^2 administered via intravenous (IV) infusion over 3 hours on Day 1 of each 21-day treatment cycle. Capecitabine 2000 mg/m^2/day was administered on Days 1 to 14 of each 21-day treatment cycle.
Period: Overall Study
Arm/Group | Ixabepilone 32 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 2000 mg/m^2/Day
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ixabepilone 40 mg/m^2 + Capecitabine 1650 mg/m^2/Day: Ixabepilone 40 mg/m^2 was administered via intravenous (IV) infusion over 3 hours on Day 1 of each 21-day treatment cycle. Capecitabine 1650 mg/m^2/day was administered on Days 1 to 14 of each 21-day treatment cycle.
- Ixabepilone 40 mg/m^2 + Capecitabine 2000 mg/m^2/Day: Ixabepilone 40 mg/m^2 was administered via intravenous (IV) infusion over 3 hours on Day 1 of each 21-day treatment cycle. Capecitabine 2000 mg/m^2/day was administered on Days 1 to 14 of each 21-day treatment cycle.
- Total: Total of all reporting groups
Arm/Group | Ixabepilone 32 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 2000 mg/m^2/Day | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 2 | 8
  >=65 years | 0 | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (13.00) | 52.7 (4.73) | 52.7 (20.26) | 53.1 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 9
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 3 | 3 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Participants Experiencing Dose Limiting Toxicity (DLT)
Description: DLT was defined as any ixabepilone and/or capecitabine related events requiring study discontinuation during the first two treatment cycles.
Time Frame: From initiation of drug through last day of Cycle 2 (Day 42)
Population: All participants who received at least 1 dose of either ixabepilone or capecitabine.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone 32 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 2000 mg/m^2/Day
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 0 | 0

2. Secondary Outcome: Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE = any new untoward medical occurrence/worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. SAE = any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event. Treatment-related=Possible, Probable, or Certain relationship to drug
Time Frame: Baseline to Day 42, continuously
Population: All participants who received at least 1 dose of either ixabepilone or capecitabine.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone 32 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 2000 mg/m^2/Day
Number analyzed (Participants) | 3 | 3 | 3
Participants
  AEs | 3 | 3 | 3
  Related AEs | 3 | 3 | 3
  Discontinued Due to AEs | 0 | 0 | 0
  SAEs | 0 | 1 | 1
  Related SAEs | 0 | 1 | 1
  Discontinued Due to SAEs | 0 | 0 | 0
  Deaths | 0 | 0 | 0

3. Secondary Outcome: Participant Tumor Response at Study Endpoint
Description: Tumor response was assessed using the Response Evaluation Criteria in Solid Tumors (RECIST) in which complete response (CR) = disappearance of all target lesions; partial response (PR) = 30% decrease in the sum of the longest diameter of target lesions; progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions; and stable disease (SD) = small changes that do not meet above criteria.
Time Frame: At baseline and after every 42 days (every 2 21-day cycles) after baseline
Population: All treated participants with measurable disease and tumor response.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone 32 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 2000 mg/m^2/Day
Number analyzed (Participants) | 3 | 3 | 3
Participants
  CR | 0 | 0 | 1
  PR | 1 | 1 | 2
  PD | 1 | 1 | 0
  SD | 1 | 1 | 0

4. Secondary Outcome: Mean Ixabepilone Maximum Plasma Concentration (Cmax) in One Dosing Interval
Description: Cmax = maximum observed plasma concentration of ixabepilone as determined from participant serum samples in one dosing interval.
Time Frame: During Cycle 1 at specified timepoints (Day 1 to Day 8).
Population: All participants who received ixabepilone and capecitabine and who had adequate PK concentration profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ixabepilone 32 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 2000 mg/m^2/Day
Number analyzed (Participants) | 3 | 3 | 3
ng/mL | 164.01 (30) | 219.44 (13) | 192.13 (6)

5. Secondary Outcome: Mean Ixabepilone Area Under the Concentration Curve (AUC INF) in One Dosing Interval
Description: AUC = the average area under the concentration curve (AUC [INF]) of ixabepilone as determined from participant serum samples in one dosing interval over 24 hours.
Time Frame: During Cycle 1 at specified timepoints (Day 1 to Day 8).
Population: All participants who received ixabepilone and capecitabine and who had adequate PK concentration profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng·h/mL
Arm/Group | Ixabepilone 32 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 2000 mg/m^2/Day
Number analyzed (Participants) | 3 | 3 | 3
ng·h/mL | 1260.71 (1) | 1676.46 (24) | 1417.78 (10)

6. Secondary Outcome: Mean Ixabepilone Terminal Elimination Half Life (T 1/2) in One Dosing Interval
Description: T 1/2 = terminal elimination half life as determined from participant serum samples in one dosing interval.
Time Frame: During Cycle 1 at specified timepoints (Day 1 to Day 8).
Population: All participants who received ixabepilone and capecitabine and who had adequate PK concentration profiles.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Ixabepilone 32 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 2000 mg/m^2/Day
Number analyzed (Participants) | 3 | 3 | 3
Hours | 41.77 (9) | 44.17 (8) | 54.27 (16)

7. Secondary Outcome: Mean Ixabepilone Volume of Distribution at Steady State (Vss) in One Dosing Interval
Description: Vss = volume of distribution at steady state determined from participant serum samples from one dosing interval.
Time Frame: During Cycle 1 at specified timepoints (Day 1 to Day 8).
Population: All participants who received ixabepilone and capecitabine and who had adequate PK concentration profiles.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Ixabepilone 32 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 2000 mg/m^2/Day
Number analyzed (Participants) | 3 | 3 | 3
Liters | 1910.13 (423) | 1498.46 (140) | 2055.55 (795)

8. Secondary Outcome: Mean Ixabepilone Total Body Clearance (CLT) in One Dosing Interval
Description: CLT = total body clearance as determined from participant serum samples in one dosing interval.
Time Frame: During Cycle 1 at specified timepoints (Day 1 to Day 8).
Population: All participants who received ixabepilone and capecitabine and who had adequate PK concentration profiles.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Ixabepilone 32 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 2000 mg/m^2/Day
Number analyzed (Participants) | 3 | 3 | 3
L/h | 41.52 (2) | 37.21 (7) | 42.79 (7)

9. Primary Outcome: Participants Achieving the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D)
Description: The MTD was defined as the highest dose evaluated for which less than 1/3 of the participants experienced DLT during the first two treatment cycles. If toxicities (e.g. hand-foot syndrome, existing peripheral neuropathy, etc.) occurred or became more severe in later cycles, the recommended Phase II dose was to be determined after due consideration of their severity.
Time Frame: At the end of Cycle 2 (Day 42)
Population: All participants treated at the highest dose level.
Measure: Number; unit: Participants
Groups:
- All Participants With Measurable Disease and Tumor Response: The evaluable participant population consisted of participants who met the minimum safety evaluation requirements of the study: participant received ≥ 1 dose of ixabepilone and/or capecitabine in Cycle 1, completed adequate safety evaluations, and was observed for ≥ 21 days following the first dose or the participant experienced DLT.
Arm/Group | All Participants With Measurable Disease and Tumor Response
Number analyzed (Participants) | 3
Participants
  Ixa 40 mg/m^2 + Cap 2000 mg/m^2 MTD | 3
  Ixa 40 mg/m^2 + Cap 2000 ng/m^2 RP2D | 3

ADVERSE EVENTS:
Groups:
- Ixabepilone 32 mg/m^2 + Capecitabine 1650 mg/m^2/Day: Ixabepilone 32 mg/m^2 was administered via intravenous (IV) infusion over 3 hours on Day 1 of each 21-day treatment cycle. Capecitabine 1650 mg/m^2/day was administered on Days 1 to 14 of each treatment cycle.
Arm/Group | Ixabepilone 32 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 1650 mg/m^2/Day | Ixabepilone 40 mg/m^2 + Capecitabine 2000 mg/m^2/Day
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone 32 mg/m^2 + Capecitabine 1650 mg/m^2/Day (N=3) | Ixabepilone 40 mg/m^2 + Capecitabine 1650 mg/m^2/Day (N=3) | Ixabepilone 40 mg/m^2 + Capecitabine 2000 mg/m^2/Day (N=3)
SKIN INFECTION (Infections and infestations) | 0 | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone 32 mg/m^2 + Capecitabine 1650 mg/m^2/Day (N=3) | Ixabepilone 40 mg/m^2 + Capecitabine 1650 mg/m^2/Day (N=3) | Ixabepilone 40 mg/m^2 + Capecitabine 2000 mg/m^2/Day (N=3)
WEIGHT DECREASED (Investigations) | 2 | 1 | 1
HAEMOGLOBIN DECREASED (Investigations) | 1 | 2 | 3
MONOCYTE COUNT DECREASED (Investigations) | 0 | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 2 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 2 | 2
FLUSHING (Vascular disorders) | 0 | 1 | 0
PHLEBITIS (Vascular disorders) | 0 | 0 | 1
SLEEP DISORDER (Psychiatric disorders) | 0 | 1 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 0 | 1
SEASONAL ALLERGY (Immune system disorders) | 0 | 0 | 1
HEADACHE (Nervous system disorders) | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 0 | 0 | 1
DYSGEUSIA (Nervous system disorders) | 0 | 1 | 2
NEURALGIA (Nervous system disorders) | 1 | 0 | 0
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 3 | 3 | 3
NAUSEA (Gastrointestinal disorders) | 1 | 3 | 2
VOMITING (Gastrointestinal disorders) | 1 | 1 | 0
CHEILITIS (Gastrointestinal disorders) | 0 | 1 | 1
DIARRHOEA (Gastrointestinal disorders) | 2 | 2 | 1
GASTRITIS (Gastrointestinal disorders) | 1 | 0 | 0
TOOTHACHE (Gastrointestinal disorders) | 0 | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 1 | 1
TONGUE PIGMENTATION (Gastrointestinal disorders) | 0 | 0 | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1 | 1
PARONYCHIA (Infections and infestations) | 1 | 1 | 1
LYMPHANGITIS (Infections and infestations) | 0 | 0 | 1
SKIN INFECTION (Infections and infestations) | 0 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 3 | 3
LEUKOPENIA (Blood and lymphatic system disorders) | 3 | 3 | 3
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 2
NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 3 | 3
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 3 | 3
RASH (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
PRURIGO (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 2 | 0 | 3
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 3 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OROPHARYNGEAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OEDEMA (General disorders) | 1 | 0 | 1
FATIGUE (General disorders) | 3 | 3 | 3
PYREXIA (General disorders) | 0 | 2 | 1
EXTRAVASATION (General disorders) | 0 | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 1
INJECTION SITE OEDEMA (General disorders) | 0 | 2 | 1
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 1 | 1
INJECTION SITE REACTION (General disorders) | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.